CLINICAL TRIAL: NCT04234607
Title: A Randomized, Double-blind, Controlled, Multicenter Phase III Study of TQB2450 or Placebo Combined With Anlotinib, Etoposide and Carboplatin Versus Etoposide and Carboplatin in Subjects With Extensive Small Cell Lung Cancer
Brief Title: A Study of TQB2450 or Placebo Combined With Anlotinib, Etoposide and Carboplatin Versus Etoposide and Carboplatin in Subjects With Extensive Small Cell Lung Cancer (ETER701)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-Ⅲ-04
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-08

CONDITIONS: Extensive Small Cell Lung Cancer
MeSH Terms: interventions — anlotinib; Etoposide; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2450+Anlotinib+ etoposide + carboplatin (Experimental): Induced stage：TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) +Etoposide (100mg/m2 IV continuously on Day 1, 2 and 3）+Carboplatin（AUC 5 mg/mL/min IV on Day 1（ maximum dosage: 800 mg）） maintenance stage：TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450; Drug: Anlotinib; Drug: Etoposide; Drug: Carboplatin
- TQB2450（blank）+Anlotinib+ etoposide + carboplatin (Experimental): Induced stage：TQB2450 (blank) 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) +Etoposide (100mg/m2 IV continuously on Day 1,2 and 3）+ Carboplatin（AUC 5 mg/mL/min IV on Day 1（ maximum dosage: 800 mg）） maintenance stage：TQB2450 (blank) 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: Anlotinib; Drug: Etoposide; Drug: Carboplatin; Drug: TQB2450（blank）
- TQB2450（blank）+Anlotinib（blank）+ etoposide + carboplatin (Active Comparator): Induced stage：TQB2450 (blank) 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib (blank) capsules 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21) +Etoposide (100mg/m2 IV continuously on Day 1,2 and 3）+Carboplatin（AUC 5 mg/mL/min IV on Day 1（ maximum dosage: 800 mg）） maintenance stage：TQB2450 (blank) 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Anlotinib capsules (blank) 12 mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: Etoposide; Drug: Carboplatin; Drug: TQB2450（blank）; Drug: Anlotinib（blank)

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: TQB2450+Anlotinib+ etoposide + carboplatin
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor
  Arms: TQB2450+Anlotinib+ etoposide + carboplatin; TQB2450（blank）+Anlotinib+ etoposide + carboplatin
Drug: Etoposide — Etoposide is a cell cycle-specific antitumor drug
Drug: Carboplatin — Carboplatin is cell cycle nonspecific antitumor drug
Drug: TQB2450（blank） — Subjects administrated TQB2450 (blank) intravenously (IV) on Day 1 of each 21-day
  Arms: TQB2450（blank）+Anlotinib+ etoposide + carboplatin; TQB2450（blank）+Anlotinib（blank）+ etoposide + carboplatin
Drug: Anlotinib（blank) — Subjects administrated anlotinib (blank) in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Arms: TQB2450（blank）+Anlotinib（blank）+ etoposide + carboplatin

SUMMARY:
A randomized, double-blind, controlled, multicenter phase III study of TQB2450 or placebo combined with Anlotinib, etoposide and carboplatin versus Etoposide and Carboplatin in subjects with extensive small cell lung cancer. The primary outcome measures include PFS and OS. Extended stage Small Cell Lung Cancer (SCLC) patients will be registered, after signing the informed consent, and then centrally randomized 1:1:1 to the experimental arms and the control arm.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed extensive small cell Lung cancer; 2. Has not received systematic treatment for extensive small cell lung cancer; 3. Has received radiotherapy and chemotherapy for limited stage SCLC must have received radical treatment, and has at least 6 months of no treatment interval from the last treatment to the diagnosis of extensive SCLC; 4. Has measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; 5. 18 and 75 years old; Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, life expectancy≥ 12 weeks; 6. Adequate organ system function; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization; 8. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has prior therapy with anlotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or other immunotherapy against PD-1/PD-L1; 2. Has central nervous system metastasis and/or cancerous meningitis; 3. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix; 4. Has multiple factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc; 5. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures; 6. Has spinal cord compression which was not cured or relieved through surgery and/or radiotherapy, or diagnosed spinal cord compression after treatment showed no clinical evidence of disease stabilization prior to randomization ≥1 week; 7. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear; 8. Within 2 months prior to initial administration, subjects with evidence or history of bleeding tendency, regardless of severity; A history of hemoptysis (defined as blood bright red or 1/2 teaspoon) or an unhealed wound, ulcer, or fracture in the 2 weeks prior to initial administration; 9. Has adverse events caused by previous therapy except alopecia that did not recover to ≤ grade 1; 10.Has major surgical procedure、biopsy or obvious traumatic injury within 28 days before randomization; 11. Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident including transient ischemic attack, deep vein thrombosis and pulmonary embolism; 12.Has drug abuse history that unable to abstain from or mental disorders; 13. Has any severe and/or uncontrolled disease; 14. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration.; 15. Severe hypersensitivity occurs after administration of other monoclonal antibodies; 16. Active autoimmune diseases requiring systemic treatment occurred within 2 years prior to first administration ; 17. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration; 18. Has participated in other anticancer drug clinical trials within 4 weeks; 19. According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 12 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 24 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) .
Disease control rate (DCR) | up to 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of response（DOR） | up to 12 months
  For participants who demonstrate CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
PFS rate of 6 and 12 months progression-free survival | up to 12 months
  PFS rate of progression-free survival at 6 and 12 months: the percentage of subjects who did not develop disease progression or die of any cause at 6 and 12 months after randomization.
OS rate of 12 and 18 months total survival | up to 12 months
  Total survival OS rate at 12 and 18 months: the proportion of subjects who died of any cause at 12 and 18 months after randomization.
Quality of life score | up to 12 months
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | up to 24 months
  Security Index

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui chest hospital, Hefei, Anhui
  - AnHui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing chest hospital，capital medical university, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Fiest Affiliated Hospital of Guanghzou University of Chinese Medicine, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Guizhou Provincial people's Hospital, Guiyang, Guizhou
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Shijiazhuang First Hospital, Shijiazhuang, Hebei
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jinzhou Central Hospital, Jinzhou, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning

REFERENCES:
- [Derived] Cheng Y, Chen J, Zhang W, Xie C, Hu Q, Zhou N, Huang C, Wei S, Sun H, Li X, Yu Y, Lai J, Yang H, Fang H, Chen H, Zhang P, Gu K, Wang Q, Shi J, Yi T, Xu X, Ye X, Wang D, Xie C, Liu C, Zheng Y, Lin D, Zhuang W, Lu P, Yu G, Li J, Gu Y, Li B, Wu R, Jiang O, Wang Z, Wu G, Lin H, Zhong D, Xu Y, Shu Y, Wu D, Chen X, Wang J, Wang M, Yang R. Benmelstobart, anlotinib and chemotherapy in extensive-stage small-cell lung cancer: a randomized phase 3 trial. Nat Med. 2024 Oct;30(10):2967-2976. doi: 10.1038/s41591-024-03132-1. Epub 2024 Jul 11. PMID 38992123